CLINICAL TRIAL: NCT05354505
Title: Fetal Endoscopic Tracheal Occlusion (FETO) Trial for Congenital Diaphragmatic Hernia (CDH)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vincent Duron (Other)
Responsible Party: Sponsor-Investigator, Vincent Duron, Associate Professor of Surgery, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAU1357
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Diaphragmatic Hernia
Keywords: Fetal Endoscopic Tracheal Occlusion (FETO); Congenital diaphragmatic hernia (CDH)
MeSH Terms: conditions — Hernia, Diaphragmatic; Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): GOLDBAL2 balloon will be placed for Fetus diagnosed with Congenital diaphragmatic hernia (CDH) at Gestational age of 27w0d - 29w6d and retrieved at Gestational age of 34w0d to 34w 6 days
  Interventions: Device: Placement of the GOLDBAL2 balloon

INTERVENTIONS:
Device: Placement of the GOLDBAL2 balloon — The Fetal Endoscopic Tracheal Occlusion (FETO) procedure using the Goldballoon Detachable Balloon (GOLDBAL2) along with the Delivery Microcatheter (BALTACCI-BDPE100) will be used to treat fetuses diagnosed with severe Congenital Diaphragmatic Hernia (CDH)

SUMMARY:
This is a single site, single arm, non-randomized, pilot trial to assess the feasibility and safety of treating severe congenital diaphragmatic hernia (CDH) with Fetal Endoscopic Tracheal Occlusion (FETO) at Columbia University Irving Medical Center (CUIMC)/ NewYork-Presbyterian Hospital (NYP).

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) affects 1 in 2,200 to 5,000 live births per year. The defect in the fetal diaphragm allows abdominal organs (intestine, stomach, liver, spleen) to migrate into the thorax, hindering normal lung development. The herniated contents place pressure on the developing lungs and this may result in varying degrees of pulmonary hypoplasia and associated pulmonary hypertension; both of which may be lethal. In an attempt to prenatally quantify the impact of the herniated organs on underlying lung development, prognostic tools have been developed. The most widely used prognostic indicator is lung-to-head ratio (LHR) as measured by prenatal ultrasound. The lung contralateral to the diaphragmatic defect is measured in a transverse plane at the level of the four chamber heart and its area is divided by the fetal head circumference (LHR). The LHR is tracked through the pregnancy but seems to be most strongly correlated with outcomes in the early third trimester.

Fetuses with severe CDH have a high risk of mortality. The current standard of care treatment offers postnatal repair, which is associated with overall survival of 71% in all cases. A majority (68%) of fetuses are prenatally diagnosed, and the survival in this cohort is even lower at 65%. The severity of the defect can be measured prenatally by the degree of pulmonary hypoplasia, and the survival drops to below 30% for those with expected lung volumes below 30% of expected. The purpose of the FETO procedure in severe CDH patients is to improve prenatal lung growth in order to potentially increase neonatal survival.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability (meets psychosocial criteria below) for the duration of the study
3. Pregnant women, age 18 years and older
4. Singleton pregnancy
5. No pathogenic variants on microarray or pathologic findings on karyotype; results by fluorescence in situ hybridization (FISH) will be acceptable if patient is >26 weeks
6. Fetal echocardiogram with changes expected with CDH and no major structural cardiac defects
7. Fetal CDH (left or right) with severe pulmonary hypoplasia, defined as o/e LHR <25% with liver up
8. Gestational age at FETO procedure: if o/e LHR <25%, will be done at 27 weeks plus 0 days to 29 weeks plus 6 days
9. Meets psychosocial criteria

   * Willing to reside within 30 minutes of NewYork-Presbyterian Sloane Hospital for Women/Columbia University Irving Medical Center (CUIMC) and ability to maintain follow up appointments. NYP/CUIMC will work with the study participant to assist in securing housing 30 minutes from the hospital if this is a challenge to her.
   * Patient has a support person (e.g. spouse, partner, friend, parent) that is available to stay with her for the duration of the pregnancy near NewYork-Presbyterian Sloane Hospital for Women/Columbia University Irving Medical Center (CUIMC)
   * Willing to comply with restrictions of daily living including inability to exercise, have intercourse, or return to work

Exclusion Criteria:

1. Multi-fetal pregnancy
2. History of latex allergy
3. History of preterm labor or incompetent cervix (requiring cerclage), short cervix (<20mm), or uterine anomaly predisposing to preterm labor
4. Psychosocial ineligibility

   * Inability to reside within 30 minutes of NewYork-Presbyterian Sloane Hospital for Women/Columbia University Irving Medical Center (CUIMC) or inability to maintain follow up appointments
   * Social work will meet with each patient to evaluate the social situation and support system. Identifiable issues of social instability or compliance with the protocol will exclude her as a potential candidate.
5. Bilateral CDH, unilateral CDH with o/e LHR > 25%, or unilateral CDH with o/e LHR <25% but liver completely down in abdomen
6. Additional fetal or genetic abnormalities that would impact care after delivery or be known to have an impact on outcome
7. Maternal contraindications to elective fetoscopic surgery
8. Significant placental abnormalities (abruption, chorioangioma, accreta) known at time of enrollment and/or surgery
9. Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy.Maternal HIV, Hepatitis B with positive surface antigen, Hepatitis C with presence of virus in maternal blood due to risk of fetal transmission during the procedure
10. No safe or feasible fetoscopic approach to balloon placement
11. Uterine anomaly such as large or multiple fibroids or mullerian duct abnormality
12. Participation in another intervention study that influences maternal and fetal morbidity and mortality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Total number of subjects with successful placement of the balloon | Up to 30 weeks
  Success will be defined as completion with direct visual placement above the carina and confirmation on ultrasound done during the procedure.
Total number of subjects with successful retrieval of the balloon | Up to 35 weeks
  Success will be defined by retrieval prior to delivery, including safe retrieval during an ex-utero intrapartum therapy (EXIT) procedure.

SECONDARY OUTCOMES:
Change in fetal lung volume growth on prenatal MRI | Baseline and up to 37 weeks
  Fetal MRI prior to balloon placement and 2nd fetal MRI at +/- 2 weeks of balloon retrieval will be performed to calculate the difference between the 1st and 2nd MRIs.
Change in fetal lung growth on prenatal ultrasound | Baseline and up to 35 weeks
  Fetal ultrasound before balloon placement and immediately prior to balloon removal will be performed to calculate the different between the 2 ultrasounds.
Gestational age at delivery | At the time of delivery (up to 40 weeks of gestation)
  Gestational age at delivery will be measured.
Total number of maternal complications | Up to 6 weeks post-delivery
  Maternal complications will be recorded and reviewed.
Survival rate post-delivery | Up to 180 days post-delivery
  Survival rate will be measured at 180 days for those still hospitalized at the time point.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Duron, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NewYork-Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No